CLINICAL TRIAL: NCT04708964
Title: Subglottic Instillation of Flurbiprofen to Prevent Laryngeal Inflammation Resulting From Endotracheal Intubation: Prospective Pilot Study, Randomized, Double Blind, Placebo Controlled.
Brief Title: Oro-tracheal Intubation: Flurbiprofen Subglottic Instillation to Prevent Laryngeal Inflammation
Acronym: SoreThroat
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.ssa M Calabrese, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sore Throat Pilot
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: D010612
Keywords: Sore Throat; Endotracheal Intubation; Flurbiprofen
MeSH Terms: conditions — Pharyngitis | interventions — Flurbiprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flurbiprofen (Active Comparator): 5 ml of flurbiprofen solution 0.25% will be administered, through the subglottic intake door of the endotracheal tube. The solution will be left in place for 1 minute
  Interventions: Drug: Flurbiprofen
- Placebo (Placebo Comparator): 5 ml of saline solution 0.9% will be administered, through the subglottic intake door of the endotracheal tube. The solution will be left in place for 1 minute
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Flurbiprofen — Flurbiprofen solution will be administered, through the subglottic intake door of the endotracheal tube.
  Arms: Flurbiprofen
Drug: saline solution — Saline solution will be administered, through the subglottic intake door of the endotracheal tube.
  Arms: Placebo

SUMMARY:
Most efficient system for airways controll during general anesthesia is oro-tracheal intubation, in order to allow mechanical ventilation and bronchial suction and to prevent gastric intake. However, in the period after exhumation, traumatism of tube placement causes in 21% to 72% of patients, sore throat (POST), generally associated hoarseness. The incidence of POST is influenced by numerous factors such as age, smoke history, duration of tube positioning maneuvers, diameter of the endotracheal tube, pressure present in the headset, duration of intubation. Although analgesics and systemically administered anti-inflammatories have been found to be effective, topical therapies based on the application of corticosteroids, NSAIDs and lidocaine are an interesting alternative because they are also effective, but devoid of the effects collateralises of systemic administration. The proposed methods for the prevention and treatment of POST in cardiac surgery patients, subjected to long-term interventions with consequent need for prolonged mechanical ventilation and therefore orotracheal intubation even in the post-operative period. The propose of trial is that the sub-glottal intake door can also be used for the peat administration of anti-inflammatory drugs in order to prevent pain caused by endotracheal intubation. This drug thus administered will directly reach the anatomical structures most involved in the genesis of post-intubation pain, that is, the vocal cords and the expected part of the trachea.

DETAILED DESCRIPTION:
Orotracheal intubation is the most efficient system for controlling the airways during general anesthesia, in order to keep them harmful, to prevent gastric intake and to allow mechanical ventilation and bronchial suction. However, a percentage ranging from 21% to 72% of patients undergoing orotracheal intubation have, in the period after exhumation, sore throat (POST) generally associated hoarseness. This complication stems from traumatism caused by tube placement and pressure exerted on the vocal cords and trachea wall during in situ parking. The incidence of POST is influenced by numerous factors such as age, smoke history, duration of tube positioning maneuvers, diameter of the endotracheal tube, pressure present in the headset, duration of intubation. The proposed methods for the prevention and treatment of POST are manifold and the literature on the subject is extensive. Several studies have assessed the effectiveness of systemic administration of opioids and NSAIDs or their peat application, by oral rinse and gargles, and the lubrication of the endotracheal tube cap with cortisonic or lidocaine-based ointments. Although analgesics and systemically administered anti-inflammatories have been found to be effective, topical therapies based on the application of corticosteroids, NSAIDs and lidocaine are an interesting alternative because they are also effective, but devoid of the effects collateralises of systemic administration. Among the drugs used in this mode there is also flurbiprofen, an NSAID successfully used in inflammation of the first airways which has also proven effective in the forms resulting from endotracheal intubation and the placement of the laryngeal mask. There are studies in the literature that have evaluated the oral administration of flurbiprofen spray. Recently, endotracheal tubes have been marketed to remove secretions that accumulate above the headset, sucking them through an accessory light. These secretions come from the upper airways and penetrate the initial part of the trachea because the presence of the endotracheal tube prevents the adduction of the vocal cords. The permanence of secretions facilitates bacterial growth and, in the long run, their passage under the cap, into the tracheobronchial tree. For this reason, the use of these tubes has been effective in reducing the incidence of pneumonia associated with invasive mechanical ventilation. The accessory light (sub-glottal suction door) has also been used to carry out washing with physiological solution, always in order to prevent material stagnation and bacterial growth above the headset. The propose of trial is that the sub-glottal intake door can also be used for the peat administration of anti-inflammatory drugs in order to prevent pain caused by endotracheal intubation. In fact, a drug thus administered will directly reach the anatomical structures most involved in the genesis of post-intubation pain, that is, the vocal cords and the expected part of the trachea. The population studied will be cardiac surgery, subjected to long-term interventions with consequent need for prolonged mechanical ventilation and therefore orotracheal intubation even in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Orotracheal intubation lasting 9-12 hours for elective interventions of myocardial revascularization or replacement/valve plastic in extracorporeal circulation and subsequent stay in intensive care.
* Ages of 50 and 75
* CLASS NYHA I or II
* Written consent to participation in the study and processing of their clinical data for the purpose of the study

Exclusion Criteria:

* Previous upper air screw surgery
* Positive history for recent acute or chronic diseases of upper airways
* Tabagism
* Positive history for difficult intubation
* Orotracheal intubation with more than two attempts or with the help of devices
* Naso-tracheal intubation
* Positive history for gastro-esophageal reflux
* Patients who have or have been affected by peptic ulcer
* Patients with known hypersensitivity (bronchial asthma, urticaria, allergic phenomena) to flurbiprofen or any of the excipients, and to aspirin and other drugs belonging to the category of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Pregnant and lactating women
* Patients participating in other experimental trials
* Patients who have not given written consent
* Any other clinical condition that the investigator says would make the patient unfit for study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of a flurbiprofen solution, administered through the subglottic intake port of endotracheal tubes, on the incidence and intensity of the Sore Throat Post Operative | ● T3: three hours after endotracheal tube removal ● T12: twelve hours after endotracheal tube removal (1 postoperative day) ● T 36: 36 hours after endotracheal tube removal (2 postoperative day) ●TDim: Time of discharge
  Decrease of Sore Throat Pain Intensity Scale (STPIS) and Throat Pain Scale (TPS)

SECONDARY OUTCOMES:
Evaluate the intensity of hoarseness Evaluate the intensity of hoarseness | ● T3: three hours after endotracheal tube removal ● T12: twelve hours after endotracheal tube removal (1 postoperative day) ● T 36: 36 hours after endotracheal tube removal (2 postoperative day) ● TDim: Time of discharge
  Categorical scale (0 = absence of hoarseness, 1= hoarseness sensation, 2= hoarseness clearly perceived by others, 3= marked hoarseness
Patients Satisfaction | ● T3: three hours after endotracheal tube removal ● T12: twelve hours after endotracheal tube removal (1 postoperative day) ● T 36: 36 hours after endotracheal tube removal (2 postoperative day) ● TDim: Time of discharge
  SATIS scale: 0 = extremely dissatisfied, 1 = very dissatisfied 2= dissatisfied 3 = a little satisfied, 4 = satisfied, 5 = very satisfied, 6 = extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Calabrese, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS

IPD SHARING:
Plan to Share IPD: No